CLINICAL TRIAL: NCT06367738
Title: Investigating the Persisting Effects of a Single Dose of Psilocybin on Structural Plasticity in Healthy Older Adults
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, Berkeley (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2024-11-14799
Record Dates: First submitted 2024-04-11; First posted 2024-04-16 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Aging
MeSH Terms: interventions — Psilocybin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Psilocybin Level 1 (Experimental): The effects of different doses of psilocybin (1 - 10 mg) will be compared.
  Interventions: Drug: Psilocybin
- Psilocybin Level 2 (Experimental): Psilocybin (11 - 20 mg) will be administered.
  Interventions: Drug: Psilocybin
- Psilocybin Level 3 (Experimental): Psilocybin (21 - 30 mg) will be administered.
  Interventions: Drug: Psilocybin

INTERVENTIONS:
Drug: Psilocybin — Psilocybin 1-30 mg

SUMMARY:
Participants in this study will undergo a series of non-invasive tests and activities designed to understand how a single dose of psilocybin might influence cognition and emotional well-being in healthy older adults. After providing written informed consent, eligible participants, aged between 60 and 85, will be randomly assigned to receive a dose of psilocybin ranging from a microdose to a moderate-to-high dose. Anatomical magnetic resonance imaging (MRI) and diffusion weighted imaging (DWI) will be used to assess changes in brain structure, while functional magnetic resonance imaging (fMRI) will be used to quantify changes in functional brain activity.

DETAILED DESCRIPTION:
The investigators will use cognitive exams, perceptual tasks, brain imaging, peripheral psychophysiology, and surveys to investigate the persisting effects of psilocybin on cognition, predictive coding, and affect in healthy older adults (60-85 years old). The investigators will measure changes in these measures by comparing baseline to one-week and one-month post-treatment. Participants will be randomly assigned to receive a dose of psilocybin in a range from microdose to moderate-to-high dose (1-30 milligrams).

Anatomical magnetic resonance imaging (MRI) and diffusion weighted imaging (DWI) will be used to assess changes in brain structure, while functional magnetic resonance imaging (fMRI) will be used to quantify changes in functional brain activity. The investigators will assess whether changes in these brain measures underlie observed changes in cognition, predictive coding and affect.

ELIGIBILITY:
Inclusion Criteria:

Are 60-85 years of age at time of Informed Consent Form signing. Are able and willing to adhere to study requirements, including attending all study visits, preparatory and follow-up sessions, and completing all study evaluations.

Are able to swallow capsules. Women of childbearing potential (WOCBP) must agree to practice an effective means of birth control throughout the duration of the study.

Have normal or corrected-to-normal vision as determined by the study staff. Written informed consent obtained from and ability for subject to comply with the requirements of the study.

Have an identified support person and agree to be accompanied home (or to an otherwise safe destination) by the support person, or another responsible party, following dosing.

Agree to inform the investigators within 48 hours of any new or changed medical conditions during the course of their study participation.

Have access to a quiet space and a computer to perform online assessments.

Exclusion Criteria:

Breastfeeding, have a positive pregnancy test at screening or at any point during the course of the study, or unwilling to practice birth control during participation in the study.

Have a current psychiatric disorder, general medical condition, or other problem or abnormality that, in the opinion of the study clinician or PI, could compromise safety, render them unsuitable for the study, or would make them unable to comply with study activities.

Have MRI contraindications (e.g., metal implants, pacemakers, claustrophobia etc.) as determined by an MRI contraindications questionnaire.

Have a history of recent, clinically significant suicidal ideation or behavior.

Have a history of a psychotic disorder, bipolar disorder (type I or II), or a dissociative disorder (determined by history).

History of Hallucinogen Persisting Perception Disorder (HPPD). History of a seizure disorder in adulthood, central nervous system (CNS) metastases or current symptomatic CNS infection.

History of intracerebral hemorrhage, embolic stroke, transient ischemic attack (TIA), or history of any aneurysmal vascular disease (including thoracic and abdominal aorta, intracranial and peripheral arterial vessels) or arteriovenous malformation.

History of valvulopathy or pulmonary hypertension. Uncontrolled hypertension (Systolic BP>139mmHG or Diastolic BP>89mmHG) or tachycardia (average HR>90bpm) averaged over at least two measurements.

Clinically significant cardiovascular disease (e.g., history of myocardial infarction or congestive heart failure); or baseline QT/QTc>500msec; or baseline QT/QTc 451-500msec with repeat QT/QTc >500msec.

Poorly controlled diabetes mellitus (e.g., history of an episode of severe hypoglycemia or hospitalization for hyperglycemia on the current diabetes regimen).

Inadequate hepatic function as determined by total bilirubin or alkaline phosphatase >3x institutional upper limit of normal; or AST or ALT >6x institutional upper limit of normal. However, participants with Gilbert syndrome are allowed to enroll.

Inadequate renal function as determined by eGFR < 30 mL/min/1.73 m2 (based on the MDRD equation) or CrCl < 30 mL/min (based on the C-G equation).

The regular use of psychotropic medications, such as antidepressants (i.e., SSRIs, tricyclic antidepressants, and monoamine oxidase inhibitors), antipsychotics, and mood stabilizers.

Concomitant dosing of psilocybin with known UGT1A10 and UGT1A9 inhibitors (e.g., diclofenac and probenecid) will be avoided. [There is no exclusion criterion based on the use of medications or substances that are inhibitors or inducers of CYP450 enzymes.]

The use of Prohibited Medications:

Serotonin Reuptake Inhibitors (SSRIs and SNRIs) Tricyclic Antidepressants (TCAs) Monoamine Oxidase Inhibitors (MAOIs) Atypical antidepressants (e.g., mirtazapine, trazodone, buspar) Antipsychotics/Neuroleptics (typical and atypical) Anti-epileptics or mood stabilizers (e.g., lithium, valproate) (does not include gabapentin used for non-epilepsy conditions) Efavirenz (Sustiva, in Atripla) Lorcaserin Over-the-counter supplements intended to affect mood or anxiety (e.g., 5HT-P, SAMe or St. John's Wort).

Other drugs associated with the serotonin syndrome (e.g., ondansetron) used within 48 hours of study drug administration.

Vasoactive drugs (e.g., sildenafil, sumatriptan, calcium channel blockers) used within 48 hours of study drug administration.

Unable to agree to the following required Lifestyle Modifications: Patients will be asked to refrain from consuming alcohol, cannabinoids, prescription analgesics/stimulants/benzodiazepines, and any recreational drugs for 48 hours before, the day of, and for 48 hours after study drug administration. Participants will be advised to consume their usual amount of coffee, tea, or other caffeine-containing beverages on the morning of their Medication Visits.

Recent and lifetime use of psychedelics (e.g. psilocybin, LSD, mescaline), entactogens (e.g. MDMA), or dissociative anesthetics (e.g. ketamine) above a predetermined threshold.

Has been diagnosed with any disease that impairs motor function (e.g., Parkinson's disease) At high risk of falls as determined by study physician considering medical history, screening of recent symptoms and medications, and functional mobility testing.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
MRI measurements of brain structure | Baseline, week 1, and week 4
  Diffusion-weighted MRI will be used to measure mean diffusivity in prefrontal cortex and hippocampus.

SECONDARY OUTCOMES:
Amplitude and pattern of fMRI cortical responses | Baseline, week 1, and week 4
  Functional magnetic resonance imaging (fMRI) responses to visual stimuli, diffusion-weighted MRI, and T1-weighted anatomical MRI will be used.
Vagus nerve reactivity | Baseline, week 1, and week 4
  Change from baseline visit on peripheral psychophysiology will be recorded using a validated task to assess vagus nerve activation during a baseline measurement compared to activation measured while viewing emotionally evocative video clips.
Perceptual measurements | Baseline, week 1, and week 4
  Perceptual measurements will be used to assess the effects of doses of psilocybin on participants' abilities to update visual prior expectations based on new information.
Penn Conditional Exclusion Test (PCET) | Baseline, week 1, and week 4
  A validated set-shifting measure of cognitive flexibility.
California Verbal Learning Test, Second Ed. (CVLT-II) | Baseline, week 1, and week 4
  A validated measure of verbal learning and memory.
Visual Reproduction (from Wechsler Memory Scale-Third Edition) | Baseline, week 1, and week 4
  A validated measure assessing ability to reproduce complex designs after a brief exposure.
Logical Memory (from Wechsler Memory Scale-Third Edition) | Baseline, week 1, and week 4
  A validated measure of recognition and recall.
Recognition memory (REC) | Baseline, week 1, and week 4
  A measurement during the in-scanner continuous MST task to assess ability to correctly distinguish between previously presented objects and novel objects.
Lure discrimination index (LDI) | Baseline, week 1, and week 4
  A measurement during the in-scanner continuous MST task to assess ability to correctly distinguish between previously presented objects and similar lure objects.
Somatic Symptom Scale-8 (SSS-8) | Baseline, week 1, and week 4
  A validated 8-item 5-point Likert scale ("not at all" to "very much") questionnaire assessing how much a subject has been bothered by various somatic symptoms in the past week such as stomach or bowel problems, feeling tired or having low energy, and headaches.
RAND 36-Item Short Form Health Survey 1.0 (SF-36, 3-items) | Baseline, week 1, and week 4
  Selected 3 items from the validated 36-item questionnaire on self-reported health. The 3 items are 6-point Likert scale and assess perceived pain in the past week and overall health.
Brief version of the Pittsburgh Sleep Quality Index (B-PSQI) | Baseline, week 1, and week 4
  A validated 6-item questionnaire assessing aspects of sleep quality in the past week.
Ryff & Keyes Psychological Wellbeing - Purpose in Life subscale (PWB-PIL) | Baseline, week 1, and week 4
  A 7-item 6-point Likert scale ("Strongly disagree" to "Strongly agree") subscale from the validated 42-item Psychological Wellbeing questionnaire. This subscale assesses the degree to which a subject perceives their life to have purpose, direction, and meaningfulness.
Social Connectedness Scale - Revised (SCS-R) | Baseline, week 1, and week 4
  A validated 20-item 6-point Likert scale ("Strongly Disagree" to "Strongly Agree") questionnaire assessing how respondents view themselves socially and the degree to which they feel socially connected with others.
Specific Emotion Experience Questionnaire (SEEQ) | Baseline, week 1, and week 4
  A 20-item 7-point Likert scale ("Not at all" to "Extremely") assessing the extent to which subjects have experienced each of the 20 listed emotions in the past week.
Big Five Inventory-2-Extra Short Form (BFI-2-XS) | Baseline, week 1, and week 4
  A validated 15-item 5-point Likert scale ("Disagree Strongly" to "Agree Strongly") questionnaire assessing various dimensions of personality. The scale has 5 dimensions: extraversion, agreeableness, conscientiousness, neuroticism, and openness.
Spontaneous Self-Distancing Questionnaire (SSDQ) | Baseline, week 1, and week 4
  A validated 2-item questionnaire assessing a subject's tendency to self-distance when reflecting on recent painful or difficult experience.
Temporal Distancing Questionnaire (TDQ) | Baseline, week 1, and week 4
  A validated 8-item 7-point Likert scale ("Does not describe me" to "Describes me extremely well") questionnaire assessing how subjects respond to negative or unpleasant life events.
Emotion Regulation Questionnaire (ERQ) | Baseline, week 1, and week 4
  A validated 10-item 7-point Likert scale ("Strongly Disagree" to "Strongly Agree") questionnaire assessing how subjects regulate and manage their emotions.
Acceptance and Action Questionnaire (AAQ-II) | Baseline, week 1, and week 4
  A validated 7-item 7-point Likert scale ("Never True" to "Always True") questionnaire assessing a subject's level of psychological flexibility and their willingness to experience difficult thoughts and emotions.
Perseverative Thinking Questionnaire (PTQ) | Baseline, week 1, and week 4
  A validated 15-item 5-point Likert scale ("Never" to "Almost always") measurement of how subjects engage with negative thoughts or problems.
Brief Resilience Scale (BRS) | Baseline, week 1, and week 4
  A validated 6-item 5-point Likert scale ("Strongly Disagree" to "Strongly Agree") self-report measure of the ability to bounce back or recover from stress.
Apathy Evaluation Scale (AES) self-rated | Baseline, week 1, and week 4
  A validated 18-item 4-point Likert scale ("not at all" to "a lot") measure of self-reported apathy.
Perceived Stress Scale (PSS) | Baseline, week 1, and week 4
  A validated 10-item 5-point Likert scale ("never" to "very often") self-report measure of perceived stress.
Supernatural Belief Scale (SBS-6) | Baseline, week 1, week 4, and week 8
  Based on the validated 10-item Supernatural Belief Scale survey to measure tendency to believe in supernatural agents, entities, and events. This 6-item version has been adapted for cross-cultural use outside of a Western Christian context. The items are on a -4 to +4 scale ("Strongly Disagree" to "Strongly Agree").
Brief Multidimensional Measure of Religiousness/Spirituality (BMMRS) | Baseline, week 1, week 4, and week 8
  A validated 40-item measure of different dimensions of religiousness and spirituality. Dimensions include: daily spiritual experiences, meaning, values/beliefs, forgiveness, private religious practices, religious and spiritual coping, religious support, religious/spiritual history, commitment, organizational religiousness, religious preference, and overall self-ranking.
Adapted version of the Credibility/Expectancy Questionnaire (CrEQ) | Week 4
  A validated 6-item measure of subjective credibility and expectation for a given intervention with 9-point Likert scale and 0%-100% (in 10% increments) questions. The language of the survey will be adapted for this intervention to focus on how subjects think the intervention will impact their well-being.
  Blinding integrity will be assessed using a multiple-choice question asking subjects to guess the dose amount that they were given
Mystical Experience Questionnaire-30 (MEQ30) | Week 4
  A validated 30-item 6-point Likert scale ("none; not at all" to "extreme [more than any other time in my life]") self-report measure of mystical-type experiences.
Challenging Experience Questionnaire (ChEQ) | Week 4
  An empirically-derived validated 26-item 6-point Likert scale of the extent to which subjects experienced challenging experiences during a psychedelic experience. The scale has 7 factors: fear, grief, physical distress, insanity, isolation, death and paranoia.
11-Dimension Altered States Questionnaire (11D-ASC) | Week 4
  A validated 56-item visual analog scale measure of multiple aspects of psychedelic experiences (e.g., Blissful state and Complex imagery) where a higher score indicates more intense subjective effects.
Persisting Effects Questionnaire - 4-item (PEQ-4) | Week 4
  A 4-item, 8-point self-report measure adapted from items developed by Griffiths et al. to assess the enduring effects of psilocybin. The 4-item version of the scale has been used in prior psilocybin trials. The items ask the participant to rate retrospectively the drug experience in terms of personal meaningfulness, spiritual significance, how psychologically challenging it was, and personal psychological insights gained. Ratings are made with respect to other life experiences (e.g., 1= "No more than routine, everyday experiences" to 8 = "The single most meaningful experience of my life")
Narrative report of subjective experience | Week 4
  Participants will write a narrative essay in response to writing prompts which will be scored using natural language processing.
Dose Estimation Scale | Week 4
  Descriptions of typical subjective experiences for the different dose amounts will be provided. Participants will then be asked to rate the certainty with which they believe they received a dose of psilocybin in that category. Certainty will be rated with a visual analog scale 0-100% where 0% is "not at all certain" and 100% is "completely certain".

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, Berkeley, Berkeley, California, United States